CLINICAL TRIAL: NCT01901107
Title: Post-Marketing Surveillance on Long-Term Drug Use of Kiklin (Bixalomer)® Capsules in Patients With Hyperphosphataemia Receiving Hemodialysis
Brief Title: Post-marketing Surveillance of Kiklin Capsules in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: KIK001
Record Dates: First submitted 2013-07-01; First posted 2013-07-17 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Renal Failure Patients With Hyperphosphataemia Receiving Hemodialysis
Keywords: Hemodialysis; CKD (chronic kidney disease); ASP1585; Hyperphosphatemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — bixalomer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Kiklin group
  Interventions: Drug: Kiklin capsules

INTERVENTIONS:
Drug: Kiklin capsules — oral
  Other Names: ASP1585; ILY101; AMG223; bixalomer

SUMMARY:
The purpose of this survey is to evaluate the safety and efficacy of long-term use of Kiklin® Capsules in actual clinical settings.

DETAILED DESCRIPTION:
Bixalomer is administered at initial oral dosage of 500 mg three times a day just before a meal. The dosage can be adjusted based on symptoms and serum phosphorus level.

ELIGIBILITY:
Chronic renal failure patients with hyperphosphataemia receiving hemodialysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic renal failure patients with hyperphosphataemia receiving hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 1078 (Actual)
Dates: Start 2013-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Safety assessed by the incidence of adverse events, physical exam and lab-tests | for one year

SECONDARY OUTCOMES:
Serum phosphate level | Baseline and 1, 2, 3, 6, 12 months after administration
Serum calcium level | Baseline and 1, 2, 3, 6, 12 months after administration
Intact PTH (parathyroid hormone) level | Baseline and 1, 2, 3, 6, 12 months after administration

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chūbu, Chubu
  - Chugoku, Chugoku
  - Hokkaido, Hokkaido
  - Kantou, Kantou
  - Kinki, Kinki
  - Kyusyu, Kyusyu
  - Shikoku, Shikoku
  - Tōhoku, Touhoku

IPD SHARING:
Plan to Share IPD: Undecided